CLINICAL TRIAL: NCT05034432
Title: Prophylactic Intra-Operative Ventricular Arrhythmia Ablation in High-Risk LVAD Candidates (PIVATAL)
Brief Title: The PIVATAL Study -Study of Ventricular Arrhythmia (VTA) Ablation in Left Ventricular Assist Device (LVAD) Patients
Acronym: PIVATAL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Huang, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00006159; R01HL159401 (NIH)
Record Dates: First submitted 2021-08-29; First posted 2021-09-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-03

CONDITIONS: Arrythmia; Cardiomyopathies
MeSH Terms: conditions — Arrhythmias, Cardiac; Cardiomyopathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-Op Prophylactic VT ablation (Experimental): Subjects will get ablation procedure as needed if they were determined to be refractory to medical antiarrhythmic control should undergo catheter-based electrophysiology study and ablation on LVAD support
  Interventions: Procedure: Intra-Op Prophylactic VT ablation
- Conventional Management (Active Comparator): To ensure uniformity in control arm, a standardized AAD regimen is recommended among subjects randomized to the medical management control arm. Subjects who are already on a stable AAD regimen, such as amiodarone, sotalol or dofetilide, these should be continued
  Interventions: Other: Conventional Management

INTERVENTIONS:
Procedure: Intra-Op Prophylactic VT ablation — For surgical intra-operative ablation, efforts will be made to identify scarred myocardium based on methods such as cardiac magnetic resonance imaging, nuclear scans, and/or echocardiogram. Electrophysiological mapping may be obtained either pre-surgery or intra-operation. Mapping and ablation will be performed with the currently approved and updated mapping and ablation systems available at each center. Voltage mapping of the ventricle(s) to delineate scars will be carried out through electroanatomic mapping
  Arms: Intra-Op Prophylactic VT ablation
Other: Conventional Management — To ensure uniformity in control arm, a standardized AAD regimen is recommended among subjects randomized to the medical management control arm. Subjects who are already on a stable AAD regimen, such as amiodarone, sotalol or dofetilide, these should be continued
  Arms: Conventional Management

SUMMARY:
To investigate the effect of VTA ablation at the time of LVAD implant to see if it can reduce the incidence of VTA after surgery

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open-label, randomized-controlled clinical trial enrolling 100 patients who are LVAD candidates with a history of VTA who will be randomized in a 1:1 ratio to intra-operative VTA ablation vs. conventional medical management. Comprehensive data on arrhythmia history, medication history will be collected in all randomized subjects. Antiarrhythmic medical therapy will be handled in a uniform pattern between the two arms. Randomized subjects will then be followed per routine schedules for post LVAD implant. Arrhythmia data, ICD therapy, additional procedures including repeat surgery, ramp echocardiographic tests, right heart catheterization and catheter-based VTA ablation will be collected. In addition, adverse events such as unplanned hospitalizations, emergency department visits, clinic visits, and all other aspects of health care utilization will be gathered. The planned average follow-up period will be 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Presence of advanced cardiomyopathy (of all INTERMACS classification) and eligible for LVAD implant per the decision of the Heart Failure clinical team
* Implanted cardioverter defibrillator (ICD) any time in past with remote monitoring or planned to undergo ICD (or ICM as an alternative, if an ICD cannot be implanted for a clinical reason) implant within the index hospitalization for LVAD implant
* History of treated or monitored sustained (i.e., >30 seconds in duration ) VT or VF episode within the past 5 years.

Exclusion Criteria:

* Past successful VTA ablation without recurrent VTA prior to LVAD implant (Patients who continue to experience VTA post ablation and pre LVAD implant qualify to be enrolled)
* Participation in other clinical trials (observational registries are allowed with approval)
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrent VTA | Post LVAD implant until end of follow-up, through study completion, an average of 18 months (minimum 6 months)
  Total VTA events, after accounting for the competing risk of death

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by medical records for hospitalization, stroke and heart failure. | Post LVAD implant until end of follow-up, approximately 18 months
  Number of participants with any of the following: hospitalization, stroke or right heart failure. Right heart failure assessed by Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) criteria.
Mean duration of LVAD implant (and ablation) surgery | Admission for LVAD implant until hospital discharge (approximately 2-4 weeks)
Mean duration of ablation | Admission for LVAD implant until hospital discharge (approximately 2-4 weeks)
Mean rate of peri-procedural complication | Admission for LVAD implant until hospital discharge (approximately 2-4 weeks)
  Peri-procedural complications include bleeding, infection, and need for repeat operation.
Mean Length of stay in the intensive care unit after LVAD implant | Admission for LVAD implant until hospital discharge (approximately 2-4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, Principal Investigator — University of Rochester
Locations (19):
- United States (19):
  - Banner University Medical Center, Phoenix, Arizona
  - UCLA Cardiac Arrthmia Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Ascension St. Vincent Indianapolis, Indianapolis, Indiana
  - Univedrsity of Louisville, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No